CLINICAL TRIAL: NCT05072899
Title: Platelet Rich Plasm Versus Hyaluronic Acid Injection in Chronic Painful Shoulder: Randomized Comparative Trial
Brief Title: Platelet Rich Plasm Versus Hyaluronic Acid Injection in Chronic Painful Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Mohamed H. ElHakeim, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Faculty of medicine Assiut uni
Record Dates: First submitted 2021-09-18; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Chronic Shoulder Pain
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 25 patient with chronic shoulder pain injected with platelet rich plasm (Experimental): patients with chronic shoulder pain injected with platelet rich plasm ultrasound guided, assessment done on initial visit and follow up after 4weeks and 6month using (VAS, CS, SPADI)
  Interventions: Procedure: platelet rich plasm
- 25 patient with chronic shoulder pain injected with Hyaluronic acid (Experimental): patients with chronic shoulder pain injected with Hyaluronic acid ultrasound guided, assessment done on initial visit and follow up after 4weeks and 6month using (VAS, CS, SPADI)
  Interventions: Procedure: Hyaluronic acid

INTERVENTIONS:
Procedure: platelet rich plasm — local injection of shoulder joint by platelet rich plasm
  Arms: 25 patient with chronic shoulder pain injected with platelet rich plasm
Procedure: Hyaluronic acid — local injection of shoulder joint by Hyaluronic acid
  Arms: 25 patient with chronic shoulder pain injected with Hyaluronic acid

SUMMARY:
Aim of This study is to compare between the effect of ultrasound-guided local injection of Platelet Rich Plasma (PRP)versus Hyaluronic (HA) for the treatment of chronic shoulder pain.

DETAILED DESCRIPTION:
This study was prospective randomized comparative trial on patients with chronic shoulder pain presented at outpatient Clinic of Physical Medicine, Rheumatology and Rehabilitation Department at Assiut University Hospitals from June 2019 to December 2020. Our study started by 70 patient with chronic shoulder pain 20 of them were missed in follow up period, the range of age from 36 - 56 years, history, clinical examination, Laboratory investigation, and imaging (X-ray or MRI) done for all patient to complete the diagnosis, patient divided randomly into two groups, Group (A) included 25 patients were treated by PRP injection and group (B) included 25 patients were treated by HA injection, both injections were performed under ultrasound (US) guidance. Randomization by sealed envelopes technique, the follow up was at the baseline, 4 weeks and 6 months post injection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age >18 years.
* Patients with chronic shoulder pain more than 6 months not responding to medical treatment or physical therapy.
* Frozen shoulder.
* Rotator cuff disorders (partial tear).

Exclusion Criteria:

* Shoulder joint instability or traumatic shoulder pain.
* Patients with local infection at the shoulder, systemic infection, or inflammatory disease (e.g., rheumatoid arthritis and hepatitis)
* Patients with a history of diabetes mellitus and malignancy (either hematological or non-hematological).
* Pregnancy.
* Patients on anticoagulant therapy.
* Injection of shoulder with corticosteroids in the preceding 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 4weeks post injection follow up.
  0-10 visual analogue scale of pain
Visual Analogue Scale (VAS) | 6 months post injection follow up
  0-10 visual analogue scale of pain
Constant score (CS) | 4weeks post injection follow up.
  This scoring system combines physical examination tests with subjective evaluations by the patients. The subjective assessment consists of 35 points and the remaining 65 points are assigned for the physical examination assessment. The subjective assessment includes a single item for pain (15 points) and 4 items for activities of daily living (20 points) (work 4, sport 4, sleep2 and positioning the hand in space 10 points). The objective assessment includes: range of motion (40 points) (forward elevation, 10 points; lateral elevation, 10 points; internal rotation, 10 points; external rotation, 10 points) and power (25 points) (scoring based on the number of pounds of pull the patient can resist in abduction to a maximum of 25 points). The total possible score is therefore 100 points.
Constant score (CS) | 6 months post injection follow up
  This scoring system combines physical examination tests with subjective evaluations by the patients. The subjective assessment consists of 35 points and the remaining 65 points are assigned for the physical examination assessment. The subjective assessment includes a single item for pain (15 points) and 4 items for activities of daily living (20 points) (work 4, sport 4, sleep2 and positioning the hand in space 10 points). The objective assessment includes: range of motion (40 points) (forward elevation, 10 points; lateral elevation, 10 points; internal rotation, 10 points; external rotation, 10 points) and power (25 points) (scoring based on the number of pounds of pull the patient can resist in abduction to a maximum of 25 points). The total possible score is therefore 100 points.
Shoulder Pain and Disability Index (SPADI) questionnaire | 4weeks post injection follow up.
  is a self-introduction administered index designed to measure the effects of different pathologic conditions on the functional status of the shoulder. All items are rated by using a visual analogue scale from "no pain" or "no difficulty" to "worst imaginable pain" or "so difficult it required help". A numerical value was obtained by dividing the scale into 11 segments from 0 to 10 for each item
Shoulder Pain and Disability Index (SPADI) questionnaire | 6 months post injection follow up
  is a self-introduction administered index designed to measure the effects of different pathologic conditions on the functional status of the shoulder. All items are rated by using a visual analogue scale from "no pain" or "no difficulty" to "worst imaginable pain" or "so difficult it required help". A numerical value was obtained by dividing the scale into 11 segments from 0 to 10 for each item

CONTACTS AND LOCATIONS:
Overall Officials: Eman H El-Hakeim, A.Professor, Principal Investigator — Assiut University-faculty of medicine
Locations (1):
- Assiut university, Asyut, Egypt